CLINICAL TRIAL: NCT00309621
Title: Safety and Efficacy of Alitretinoin in the Treatment of Severe Refractory Chronic Hand Dermatitis
Brief Title: Safety and Efficacy of a Retinoid for the Treatment of Severe Chronic Hand Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAP00626
Record Dates: First submitted 2006-03-30; First posted 2006-04-03 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Hand Dermatoses
Keywords: Hand Dermatoses,; hand dermatitis; hand eczema; chronic hand dermatitis; retinoid
MeSH Terms: conditions — Hand Dermatoses | interventions — Alitretinoin

INTERVENTIONS:
Drug: alitretinoin

SUMMARY:
Patients with severe chronic hand dermatitis, that has not responded to topical treatment, including topical steroids and the avoidance of aggravating factors, will be treated with the oral medication alitretinoin. The study aims to investigate the safety and efficacy of the medication when given over a period of 6 months.

DETAILED DESCRIPTION:
For severe, chronic hand dermatitis, refractory to topical treatment and the avoidance of aggravating factors such as allergens and irritants, no registered systemic treatment is available. Current systemic treatment options consist in the off-label use of systemic immune suppressants, such as cyclosporine, methotrexate.

Severe chronic hand dermatitis is a debilitating disease, with massive impact on social life and working ability. A huge proportion of the population suffers for more than a decade, and job losses are a frequent consequence.

This open-label trial investigates the safety and efficacy of oral alitretinoin 30mg as a single daily dose for up to 6 months. The trial is complementary to the pivotal efficacy study BAP00089.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hand dermatitis, rated as severe by physicians global assessment, present for at least 6 months, that has not responded to the avoidance of allergens and irritants and the use of topical steroids

Exclusion Criteria:

* female of childbearing potential, unless participating in a pregnancy prevention program
* psoriasis
* active major psychiatric condition

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2006-04; Primary Completion 2007-04 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Safety:
Adverse Events
Safety Laboratory
Radiological investigations (bone density, x-ray)

SECONDARY OUTCOMES:
Physicians Global Assessment
modified Total Lesion Symptom Score
Patients Global Assessment
Patient Defined Outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Diepgen, MD, Principal Investigator — Univ. Heidelberg
Locations (30):
- Canada (10):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Hawkesbury, Ontario
  - London, Ontario
  - Markham, Ontario
  - Oakville, Ontario
  - Montreal, Quebec
  - Sheerbroke, Quebec
  - Québec
- Germany (14):
  - Berlin
  - Cologne
  - Frankfurt
  - Hamburg
  - Abt. Klinische Sozialmedizin, Heidelberg
  - Ibbenbueren
  - Lübeck
  - Mönchengladbach
  - München
  - Münster
  - Osnabrück
  - Potsdam
  - Viersen
  - Wuppertal
- Poland (6):
  - Gdansk
  - Krakow
  - Lublin
  - Opole
  - Szcecin
  - Wroclaw

REFERENCES:
- [Background] Ruzicka T, Larsen FG, Galewicz D, Horvath A, Coenraads PJ, Thestrup-Pedersen K, Ortonne JP, Zouboulis CC, Harsch M, Brown TC, Zultak M. Oral alitretinoin (9-cis-retinoic acid) therapy for chronic hand dermatitis in patients refractory to standard therapy: results of a randomized, double-blind, placebo-controlled, multicenter trial. Arch Dermatol. 2004 Dec;140(12):1453-9. doi: 10.1001/archderm.140.12.1453. PMID 15611422
- [Derived] Blome C, Maares J, Diepgen T, Jeffrustenbach S, Augustin M. Measurement of patient-relevant benefits in the treatment of chronic hand eczema--a novel approach. Contact Dermatitis. 2009 Jul;61(1):39-45. doi: 10.1111/j.1600-0536.2009.01536.x. PMID 19659963